CLINICAL TRIAL: NCT02907710
Title: A Multicenter, Prospective, Randomized Controlled Clinical Trial Comparing Endostar With Concurrent Chemoradiotherapy and Concurrent Chemoradiotherapy in the Treatment of Locoregionally Advanced Nasopharyngeal Carcinoma (NPC)
Brief Title: Endostar Combined With Concurrent Chemoradiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, min kang, doctor, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstGuangxiMU
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; endostar; chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — endostar protein; Endostatins

ARMS (2):
- concurrent chemoradiotherapy + endostar (Experimental): Drug: Endostar
  Endostar 7.5mg / m2,3 cycles of intravenous infusion for ten days, and 2 cycles of maintenance therapy after radiotherapy
  Drug: DDP
  DDP 100mg / m2, intravenous infusion over 2 hours , for 2-3 cycles
  Radiation: IMRT
  IMRT:70-74Gy
  Interventions: Drug: Endostar; Drug: DDP
- concurrent chemoradiotherapy (Active Comparator): Drug: DDP
  DDP 100mg / m2, intravenous infusion over 2 hours , for 2-3 cycles
  Radiation: IMRT
  IMRT:70-74Gy
  Interventions: Drug: DDP

INTERVENTIONS:
Drug: Endostar — intravenous infusion
  Other Names: recombinant human endostatin
  Arms: concurrent chemoradiotherapy + endostar
Drug: DDP

SUMMARY:
A total of 300 patients with pathologically confirmed Locoregionally advanced nasopharyngeal carcinoma were enrolled. Patients were randomly divided into two groups, with 150 patients in each group. One group was treated with Concurrent Chemoradiotherapy combined with Endostar and the other group was treated with Concurrent Chemoradiotherapy. The short term efficacy and the toxic and side effects of these treatments were evaluated. The 1-year, 3-year, 5-year overall survival and progression-free survival of patients were analyzed. The investigators data may provide an alternative option for the treatment of Locoregionally advanced nasopharyngeal carcinoma with high efficacy and low toxicity.

DETAILED DESCRIPTION:
This study was a multicenter, prospective, randomized controlled clinical trial. A set of unified standards were used, including the clinical research program, inclusion criteria, exclusion criteria, chemoradiotherapy regimen and evaluation criteria. Five medical centers participated in this study and 300 patients with pathologically confirmed Locoregionally advanced nasopharyngeal carcinoma were enrolled. These patients were stratified according to clinical stage and participating center, and were randomly divided into two groups: concurrent chemoradiotherapy combined with Endostar group ( IMRT 70-74Gy, Endostar 7.5mg / m2, 3 cycles of intravenous infusion, and 2 cycles of maintenance therapy after radiotherapy) and concurrent chemoradiotherapy group ( IMRT 70-74Gy, DDP 100mg / m2, intravenous infusion over 2 hours , for 2-3 cycles). After treatment, follow-up was performed every 3 months. The treatment toxicity, local control rate, distant metastasis-free survival, overall survival, progression-free survival were observed and assessed.

ELIGIBILITY:
Inclusion Criteria:

1. patients of either gender and aged from 18 to 70 years old.
2. patients with histologically confirmed non-keratinizing squamous cell nasopharyngeal carcinoma.
3. patients at stage III/IVb by UICC2010 staging.
4. KPS ≥ 70 (Appendix I)
5. patients with available MRI data of nasopharynx and measurable tumor lesions.
6. patients did not receive any treatment before enrollment.
7. patients with expected survival longer than 6 months.
8. biochemical indexes: hemoglobin > 120 g/L, WBC > 4 x 109 /L, and blood platelet ≥ 100 x 109 /L; levels of indicators for hepatic and renal function was 1.25 folds of the upper limit of normal value.
9. the informed content was obtained from every patient.
10. patients with effective follow-up.

Exclusion Criteria:

1. those with malignant tumors other than nasopharyngeal carcinoma, stage I non-melanoma skin cancer, and cervical carcinoma in situ.
2. those received treatments before enrollment.
3. pregnant or lactating women and reproductive women without contraception.
4. those who were undergoing other drug trials.
5. those with severe complications, including myocardial infarction, severe arrhythmia, severe cerebrovascular disease, ulcer disease, mental illness and uncontrollable diabetes.
6. those who could not be followed up at regular intervals.
7. those who were treated with tumor targeting drugs.
8. those who could not subject to MRI examination.
9. those who could not meet the requirements of the prescribed dose.
10. those with hemorrhagic tendency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
3-year Progression Free Survival | 3 years
  The subjects were randomly divided into two groups. Group A: concurrent chemoradiotherapy combined with Endostar，including 3 cycles of intravenous infusion, and 2 cycles of maintenance therapy after radiotherapy，and Group B: concurrent chemoradiotherapy, concurrent chemotherapy for 2 or 3 cycles. After treatment, the subjects go into observation period. MRI will be used for evaluating the carcinoma status. During 3 years, any relapse or death will be recorded.

SECONDARY OUTCOMES:
5-year Overall Survival | 5 years
  The subjects were randomly divided into two groups. Group A: concurrent chemoradiotherapy combined with Endostar，including 3 cycles of intravenous infusion, and 2 cycles of maintenance therapy after radiotherapy，and Group B: concurrent chemoradiotherapy, concurrent chemotherapy for 2 or 3 cycles. After treatment, the subjects go to observation period for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: sheng ren wang, doctor, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Result] Lee AW, Sze WM, Au JS, Leung SF, Leung TW, Chua DT, Zee BC, Law SC, Teo PM, Tung SY, Kwong DL, Lau WH. Treatment results for nasopharyngeal carcinoma in the modern era: the Hong Kong experience. Int J Radiat Oncol Biol Phys. 2005 Mar 15;61(4):1107-16. doi: 10.1016/j.ijrobp.2004.07.702. PMID 15752890
- [Result] Lee N, Harris J, Garden AS, Straube W, Glisson B, Xia P, Bosch W, Morrison WH, Quivey J, Thorstad W, Jones C, Ang KK. Intensity-modulated radiation therapy with or without chemotherapy for nasopharyngeal carcinoma: radiation therapy oncology group phase II trial 0225. J Clin Oncol. 2009 Aug 1;27(22):3684-90. doi: 10.1200/JCO.2008.19.9109. Epub 2009 Jun 29. PMID 19564532
- [Result] Kyzas PA, Cunha IW, Ioannidis JP. Prognostic significance of vascular endothelial growth factor immunohistochemical expression in head and neck squamous cell carcinoma: a meta-analysis. Clin Cancer Res. 2005 Feb 15;11(4):1434-40. doi: 10.1158/1078-0432.CCR-04-1870. PMID 15746043
- [Result] Qian CN, Zhang CQ, Guo X, Hong MH, Cao SM, Mai WY, Min HQ, Zeng YX. Elevation of serum vascular endothelial growth factor in male patients with metastatic nasopharyngeal carcinoma. Cancer. 2000 Jan 15;88(2):255-61. PMID 10640954
- [Result] Krishna SM, James S, Balaram P. Expression of VEGF as prognosticator in primary nasopharyngeal cancer and its relation to EBV status. Virus Res. 2006 Jan;115(1):85-90. doi: 10.1016/j.virusres.2005.07.010. Epub 2005 Sep 1. PMID 16139912
- [Result] Druzgal CH, Chen Z, Yeh NT, Thomas GR, Ondrey FG, Duffey DC, Vilela RJ, Ende K, McCullagh L, Rudy SF, Muir C, Herscher LL, Morris JC, Albert PS, Van Waes C. A pilot study of longitudinal serum cytokine and angiogenesis factor levels as markers of therapeutic response and survival in patients with head and neck squamous cell carcinoma. Head Neck. 2005 Sep;27(9):771-84. doi: 10.1002/hed.20246. PMID 15920746
- [Result] Huang X, Wong MK, Zhao Q, Zhu Z, Wang KZ, Huang N, Ye C, Gorelik E, Li M. Soluble recombinant endostatin purified from Escherichia coli: antiangiogenic activity and antitumor effect. Cancer Res. 2001 Jan 15;61(2):478-81. PMID 11212235